CLINICAL TRIAL: NCT02258282
Title: Safety and Efficacy of Etanercept in Patients With Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YSP20140688
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept (Experimental): Patients under the treatment of 50 mg Etanercept
  Interventions: Drug: Etanercept
- Control (Sham Comparator): Patients under the treatment of traditional DMARDs
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Etanercept
  Arms: Etanercept
Drug: Control
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of etanercept in patients with psoriasis who had an unsatisfactory response to traditional DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* has plaque psoriasis and has shown an unsatisfactory response to traditional DMARDs
* 18 to 75 years old
* has PGA of 3 or more at Day 0
* has BSA of 3% or more at Day 0
* has psoriasis severe enough to be eligible to systemic therapy
* willing to use an effective method of contraception for at least 30 days before Day 0 and until at least 1 month after the last drug administration;
* capable of giving informed consent
* with normal or non clinically significant chest X-ray within 6 months prior to Day 0
* with negative Purified Protein Derivative (PPD) or Quantiferon TB Gold test within 90 days prior to Day 0
* female patients of childbearing potential have a negative serum pregnancy test
* patient is able to start etanercept per the approved product monograph

Exclusion Criteria:

* has used topical steroids, topical tar preparations, or other anti-psoriatic preparations within the two weeks prior to Day 0 or during the study period
* has presence of erythrodermic, pustular or guttate psoriasis
* has had significant infections within the 30 days prior to Day 0
* has received investigational drugs within the four weeks prior to screening or during the study period
* has been treated with systemic anti-psoriatic drugs such as steroids, retinoids, cyclosporine, PUVA therapy or methotrexate within the four weeks prior to Day 0 or during the study period
* received systemic antibiotics within the four weeks prior to Day 0
* has been treated with ultraviolet light therapy (UVB, nbUVB) within the two weeks prior to Day 0 or during the study period
* has used infliximab within 14 days of Day 0 or during the study period
* has used other biologic agents for the treatment of psoriasis besides etanercept 8 weeks prior to Day 0 or during the study period
* has had an allergic reaction to infliximab
* has an unstable or serious medical condition as defined by the investigator or presence of any significant medical condition that might cause this study to be detrimental to the patient
* uncontrolled or severe comorbidities such as poorly controlled diabetes mellitus, NYHA class III or IV heart failure, history of myocardial infarction or cerebrovascular accident or transient ischemic attack within three months of screening visit; unstable angina pectoris
* uncontrolled hypertension, oxygen-dependent severe pulmonary disease
* has a known sero-positivity for HIV virus or history of any other immunosuppressive disease
* has active or chronic Hepatitis B or C
* has any mycobacterial disease, patient with a chest X-Ray suggestive of tuberculosis or patient taking anti-tuberculosis medication
* has a known hypersensitivity to etanercept or one of its components
* has received a live attenuated vaccine within the 12 weeks prior to Day 0 or plans to receive one during the study
* current pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-05; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of Physician's Global Assessment (PGA) at 24 weeks | At 0 week, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Mean Body Surface Area (BSA) | At 0 week, 12 weeks, 24 weeks
Mean Psoriasis Area and Severity Index (PASI) | At 0 week, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chengdu Military Area Command PLA, Chengdu, Sichuan, China